CLINICAL TRIAL: NCT01444131
Title: A 26-Week Phase II, Multicentre, Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Varenicline in Combination With Nicotine Replacement Therapy for Smoking Cessation
Brief Title: Varenicline in Combination With Nicotine Replacement Therapy for Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Collaborators: QuitSupport (Unknown)
Responsible Party: Principal Investigator, Prof Elvis M Irusen, Clinical Professor, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VarNic
Record Dates: First submitted 2011-09-27; First posted 2011-09-30 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Tobacco Dependence
Keywords: Smoking; Smoking cessation; Pharmaceutical aids
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation | interventions — Varenicline; Tobacco Use Cessation Devices; Nicotine Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline and Placebo Patch (Placebo Comparator): Varenicline and Nicotine Patch (placebo)
  Interventions: Drug: Varenicline and Placebo Patch
- Varenicline and Nicotine Patch (Active Comparator): Varenicline and Nicotine Patch 15mg
  Interventions: Drug: Varenicline, Nicotine Patch

INTERVENTIONS:
Drug: Varenicline, Nicotine Patch — active nicotine patches added to varenicline.
  Other Names: Champix; Nicorette
  Arms: Varenicline and Nicotine Patch
Drug: Varenicline and Placebo Patch — placebo nicotine patches added to varenicline.
  Arms: Varenicline and Placebo Patch

SUMMARY:
The purpose of this study is to test whether the addition of a nicotine patch to varenicline increases smoking cessation success rate and whether the combination is safe.

DETAILED DESCRIPTION:
This is a phase-II multicenter study involving 438 smokers, to be conducted at 7 sites in South Africa, over 6 months. In a randomized 1:1 allocation varenicline tartrate 1 mg twice daily, given in an incremental dosage for the first week before target quit date (TQD), will be compared to varenicline tartrate in the same dose combined with a 15mg nicotine patch. The nicotine patch (active and placebo) will be provided by McNeil. The patch will be given 2 weeks prior TQD. Treatment duration from TQD is 12 weeks with varenicline being tapered off during week 13.

A total of 12 clinic visits and 1 telephonic contact is planned for the 6-month study duration. The main efficacy outcome will be the 4-week continuous abstinence rate during the last four weeks of treatment, i.e. weeks 9 - 12. Efficacy assessments will be based on a Nicotine Use Inventory and measurements of end-expiratory exhaled carbon monoxide. Safety assessments will be based on adverse events evaluation, with special attention being given to the occurrence of nausea during the pretreatment period, as well as neuro-psychiatric symptoms such as depression or suicidal ideation. Participants will not be subjected to any invasive procedures.

This protocol is based on current evidence and two further abstracts presented at the European Respiratory Society Conference in Vienna, September 2009, that a combination of varenicline tartrate and nicotine replacement therapy indicate superior efficacy in cessation rate, but also an excellent good safety profile.

This study relates to the area of pharmacotherapy of smoking cessation, and will answer a frequently asked question. Importantly, several leading pulmonologists with experience in smoking cessation in South Africa have expressed their keen interest to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Current cigarette smokers, male and female, aged between 18-75 years (both limits inclusive), and who are motivated to stop smoking.
2. Have smoked on average at least 10 cigarettes per day during past year and during the month prior to screening, and no period of abstinence greater than 3 months in the past year.
3. Women of child-bearing potential (WCBP) may be included provided they are not pregnant, not nursing, and meet all of the following criteria:

   * instructed and agree to avoid pregnancy through 30 days after the last dose of study medication
   * negative screening test (beta-HCG) at screening
   * agree to use at least one birth control method (oral contraceptive, IUD, implantable or injectable contraceptive for at least 1 month prior to entering the study and will continue its use through at least 30 days after the last dose of study medication, or use a barrier method of contraception (p.e.condom, diaphragm with spermicide) while participating in the study through at least 30 days after the last dose of study medication; or abstinence.
4. Patients must have no serious or unstable disease in the past 6 months.
5. Patients must be able to be outpatients, to be assessed in a clinical setting, and be able and willing to comply with all study visits during the treatment and non-treatment periods.
6. Only one subject per household may participate.

Exclusion Criteria:

1. Patients currently suffering from depression or who have been diagnosed with depression or treated with anti-depressants within the past 12 months.
2. Patients with a past of present history of psychosis, panic disorder, or bipolar disorder.
3. Patients with severe chronic obstructive pulmonary disease (COPD).
4. Patients with clinically significant cardiovascular disease in the past 6 months. such as myocardial infarction, coronary artery bypass graft (CABG), percutaneous transluminal coronary angioplasty (PTCA), severe or unstable angina, serious arrhythmia, and clinically significant ECG conduction abnormalities.
5. Patients with uncontrolled hypertension or a systolic blood pressure greater than 150mmHg or as diastolic pressure greater than 95mmHg at screening or baseline.
6. Patients with clinically significant neurological disorders or cerebrovascular diseases (for example, stroke, transient ischemic attack, etc.) in the past 6 months.
7. Patients with a history of clinically significant endocrine disorders or gastrointestinal diseases, including insulin dependent diabetes mellitus, uncontrolled hyperthyroidism, and active peptic ulcer.
8. Patients with clinically significant hepatic or renal impairment or other clinically significant abnormal laboratory test values.
9. Patients with a history of cancer (cured basal cell or squamous cell carcinoma of the skin allowed).
10. Patients with a history of clinically significant allergic reactions to drugs (for example, severe cutaneous and/or systemic allergic reactions).
11. Patients with a history of drug (except nicotine) or alcohol abuse or dependence within the past 12 months.
12. Patients with a body mass index (BMI) less than 15 or greater than 38 when wearing indoor clothing without shoes. No subject will be enrolled with a weight less than 45.5kg (100 pounds).
13. Patients previously enrolled in a study that included varenicline.
14. Patients having used nicotine replacement therapy within the last 6 months.
15. Patients taking another investigational drug within 30 days or 5 half-lives (whichever is longer) before the Baseline visit or within 30 days of study completion.
16. Use of prohibited medications: any antidepressants, including bupropion; antipsychotic agents; mood stabilizers; naltrexone; steroids (inhaled and topical steroids are permitted); insulin.
17. Patients who do not agree to completely abstain from using non-cigarette tobacco products (including for example, pipe tobacco, cigars, snuff, chewing tobacco, etc.) or marijuana during study participation.
18. Patients who intend to donate blood or blood components while receiving study drug or within 1 month of the completion of the study treatment.
19. Patients unable/or unlikely to comprehend and follow the study protocol, including patients unable and/or unwilling to participate in the non-treatment follow-up. Patients who, in the investigator's opinion, will be unlikely to commit to a 6 month-long study.
20. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
continuous abstinence (CAR) from weeks 9 to 12 of treatment | 3 months
  The primary endpoint is the 4-week continuous abstincence rate for week 9 - 12 of treatment, i.e. the proportion of patients who are able to maintain complete abstinence from cigarette smoking and other nicotine use, with end-expiratory exhaled carbon monoxide (CO) measurements 10 ppm or less, for the planned last 4 weeks of treatment.

SECONDARY OUTCOMES:
CAR from weeks 9 to 24 | 6 months
  The secondary endpoint is the 4-week continuous abstincence rate for week 9 - 24 of treatment, i.e. the proportion of patients who are able to maintain complete abstinence from cigarette smoking and other nicotine use, with end-expiratory exhaled carbon monoxide (CO) measurements 10 ppm or less, for the planned last 4 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Elvis M Irusen, MBChB, FCP, PhD, Principal Investigator — University of Stellenbosch
Locations (7):
- South Africa (7):
  - Respiratory Research Unit, Cape Town, Western Cape
  - Synopsis Research, Cape Town, Western Cape
  - UCT Lung Institute, Cape Town, Western Cape
  - Dr JA O'Brien, Cape Town, Western Cape
  - Dr AHH Brüning, Gatesville / Cape Town, Western Cape
  - Dr MS Abdool-Gaffar, eManzimtoti
  - Dr C Smith, Sandton

REFERENCES:
- [Background] Gonzales D, Rennard SI, Nides M, Oncken C, Azoulay S, Billing CB, Watsky EJ, Gong J, Williams KE, Reeves KR; Varenicline Phase 3 Study Group. Varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs sustained-release bupropion and placebo for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):47-55. doi: 10.1001/jama.296.1.47. PMID 16820546
- [Background] Jorenby DE, Hays JT, Rigotti NA, Azoulay S, Watsky EJ, Williams KE, Billing CB, Gong J, Reeves KR; Varenicline Phase 3 Study Group. Efficacy of varenicline, an alpha4beta2 nicotinic acetylcholine receptor partial agonist, vs placebo or sustained-release bupropion for smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):56-63. doi: 10.1001/jama.296.1.56. PMID 16820547
- [Background] Tonstad S, Tonnesen P, Hajek P, Williams KE, Billing CB, Reeves KR; Varenicline Phase 3 Study Group. Effect of maintenance therapy with varenicline on smoking cessation: a randomized controlled trial. JAMA. 2006 Jul 5;296(1):64-71. doi: 10.1001/jama.296.1.64. PMID 16820548
- [Background] Tonnesen P, Paoletti P, Gustavsson G, Russell MA, Saracci R, Gulsvik A, Rijcken B, Sawe U. Higher dosage nicotine patches increase one-year smoking cessation rates: results from the European CEASE trial. Collaborative European Anti-Smoking Evaluation. European Respiratory Society. Eur Respir J. 1999 Feb;13(2):238-46. doi: 10.1034/j.1399-3003.1999.13b04.x. PMID 10065662
- [Background] Schuurmans MM, Diacon AH, van Biljon X, Bolliger CT. Effect of pre-treatment with nicotine patch on withdrawal symptoms and abstinence rates in smokers subsequently quitting with the nicotine patch: a randomized controlled trial. Addiction. 2004 May;99(5):634-40. doi: 10.1111/j.1360-0443.2004.00711.x. PMID 15078238
- [Background] Shiffman S, Ferguson SG. Nicotine patch therapy prior to quitting smoking: a meta-analysis. Addiction. 2008 Apr;103(4):557-63. doi: 10.1111/j.1360-0443.2008.02138.x. PMID 18339101
- [Background] Bolliger CT, Zellweger JP, Danielsson T, van Biljon X, Robidou A, Westin A, Perruchoud AP, Sawe U. Smoking reduction with oral nicotine inhalers: double blind, randomised clinical trial of efficacy and safety. BMJ. 2000 Aug 5;321(7257):329-33. doi: 10.1136/bmj.321.7257.329. PMID 10926587
- [Background] Ebbert JO, Burke MV, Hays JT, Hurt RD. Combination treatment with varenicline and nicotine replacement therapy. Nicotine Tob Res. 2009 May;11(5):572-6. doi: 10.1093/ntr/ntp042. Epub 2009 Apr 7. PMID 19351781
- [Background] Bolliger CT, van Biljon X, Axelsson A. A nicotine mouth spray for smoking cessation: a pilot study of preference, safety and efficacy. Respiration. 2007;74(2):196-201. doi: 10.1159/000097136. Epub 2006 Nov 14. PMID 17108670
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Koegelenberg CF, Noor F, Bateman ED, van Zyl-Smit RN, Bruning A, O'Brien JA, Smith C, Abdool-Gaffar MS, Emanuel S, Esterhuizen TM, Irusen EM. Efficacy of varenicline combined with nicotine replacement therapy vs varenicline alone for smoking cessation: a randomized clinical trial. JAMA. 2014 Jul;312(2):155-61. doi: 10.1001/jama.2014.7195. PMID 25005652